CLINICAL TRIAL: NCT03658239
Title: The Investigation of Corneal Biomechanics Through the Changes in the Intraocular Pressure
Brief Title: Corneal Biomechanics Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational Issues.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Geunyoung Yoon, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 71844
Record Dates: First submitted 2018-06-01; First posted 2018-09-05 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Subjects will undergo 4-5 visits total over the course of 6 months. There will be 3-4 visits that will be done at the Flaum Eye Institute. During these sessions the subject will be measured with a stationary topographer (GALILEI G4), with a rotatable topography measurement (Oculus Topographer) and a Tonometer. The subject's heart rate and blood pressure will also be measured (using a commercially available blood pressure and heart rate meter).
  The GALILEI measurement will only be done once. The rest of the measurements will be done up to 4 times. Once at the start of the study session then, after the subject has been inverted using a commercially available inversion table to first 135 degrees, then 150 degrees and finally to 165 degrees.
  The blood pressure and heart rate will be monitored to ensure subject safety.
  There will also be one visit at the Massachusetts General Hospital. The visit will be 2 hours and will involve a Brillouin Microscopy measurement.
  Interventions: Other: Inversion

INTERVENTIONS:
Other: Inversion — Inversions will be done while the subject is on the inversion table. The subject will be inverted to 135, 150 and 165 degrees. There inversion will not last longer than 3 minutes at a time. The inversion will be terminated if the subject's blood pressure drops below 50 mmHg diastolic or if the subject's blood pressure increases more than 50 mmHg systolic.

SUMMARY:
The goal of the study is to investigate relationship between the corneal response to a temporary increase in intraocular pressure and corneal mechanical properties.

DETAILED DESCRIPTION:
The preliminary theoretical study in which the corneal geometry at different intraocular pressure (IOP) levels is investigated using a theoretical biomechanical cornea model found changes in both conventional refractive error (sphere and cylinder) and irregular astigmatism i.e. higher order aberrations (e.g. spherical aberration, trefoil and quadrafoil). This is due to the mechanical characteristics of the cornea determined largely by interaction between collagen fibrils organization and extrafibrillar matrix material properties. Corneal geometry and the material properties are the two main factors that contribute to the changes in corneal aberrations with IOP elevation. These aberration changes due to the variation of IOP and the material properties of the cornea can be measured routinely with corneal topography systems (UR) and Brillouin ocular scanner (MGH), respectively and can guide the investigators to study their impact on optical and biomechanical behaviors of the cornea.

ELIGIBILITY:
Inclusion Criteria

A person is eligible for inclusion in the study if he/she:

* Is an adult between the ages of 18 and 55.
* Is under 250 pounds.

Exclusion Criteria

A person will be excluded from the study if he/she:

* Is under the age of 18 or over the age of 55 yrs.
* Weighs more than 250 pounds.
* Has clinically significant dry eye.
* Has glaucoma.
* Has hypertension.
* Has prior CVA.
* Has cardiovascular disease.
* Has lower extremity joint injury, damage, or replacement.
* Has baseline bradycardia.
* Has any orthopaedic injuries.
* Is pregnant.
* Has hiatal and ventral hernias.
* Has vertigo.
* Has acid reflux (GERD).
* Is undergoing myopia control treatment (e.g. atropinisation, Ortho-K, bifocal contact lenses etc.).
* Has conditions or has undergone procedures resulting in significant corneal irregularity (e.g. keratoconus, corneal transplant, etc.). This does not include astigmatism and basic refractive errors.
* Has any ocular or systemic diseases that, in the opinion of the PI/SI, would interfere with obtaining a measurement.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Corneal Surface Topography Measurement | 6 months
  Corneal Surface Topography measurement will be collected at each of the 3-4 study visits at the Flaum Eye Institute. The numerical data generated will be analyzed and compared within each subject as well as across subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Geunyoung Yoon, PhD, Principal Investigator — University of Rochester

IPD SHARING:
Plan to Share IPD: No